CLINICAL TRIAL: NCT02644044
Title: Intrathecal Methotrexate for Progressive Multiple Sclerosis: An Open Label Single Arm Study
Acronym: ITMTXPMS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director R&D Division, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0166-15-TLV
Record Dates: First submitted 2015-03-23; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: To Evaluate the Effect of Therapy With IT MTX on the Disease Course of Patients With Progressive MS
Keywords: Progressive multiple sclerosis; methotrexate
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Treatment with IT methotrexate
  Interventions: Drug: Intrathecal methotrexate

INTERVENTIONS:
Drug: Intrathecal methotrexate — 12.5 mg of methotrexate diluted to a concentration of up to 4 mg/mL in 0.9 percent sodium chloride with 4 mg Dexamethasone via lumbar puncture needle.

SUMMARY:
Multiple sclerosis (MS) is characterized pathologically by demyelination, axonal loss, and glial scar formation. Clinically, most patients have a relapsing-remitting course of MS (RRMS) that over time may become progressive without remissions - a secondary progressive MS (SPMS). About 15% of patients have a progressive course from onset which is called primary progressive (PP).

Currently, there is no approved treatment for PPMS and for SPMS only therapy with mitoxantrone showed mild effect. Thus, more effective therapies need to be developed for treatment of SPMS and PPMS.

Methotrexate (MTX), an anti-metabolite, has been in clinical use since 1948 when it was found to produce temporary remission of acute childhood leukemia.

There are accumulating evidences that in progressive MS patients there are follicular lymphoid structures in the meninges and in the Virchow-Robin spaces. Therefore, intrathecal therapy may target the pathological follicular lymphoid activity.

The safety of intrathecal MTX (ITMTX) has been demonstrated by its widespread use in treating lymphoproliferative diseases and leptomeningeal metastases. Sadik et. Al. reported about the feasibility and safety of using intrathecal methotrexate (ITMTX) as a treatment for unresponsive patients with progressive forms of MS. In their open label study they found that ITMTX may have a beneficial effect in progressive forms of MS and that it was well tolerated with no serious adverse events.

The investigators aim is to evaluate the efficacy , safety and tolerability of intrathecal methotrexate administration every 3 months in progressive 30 patients with progressive MS. The investigators will evaluate clinical, laboratory evaluation of the blood and cerebrospinal fluid as well as the MRI scans of the participants. Each patient will be treated 4 times for 1 year with the option to continue for another 1 more year with the same protocol.

DETAILED DESCRIPTION:
Protocol Intrathecal Methotrexate for Progressive Multiple Sclerosis: An Open Label Single Arm Study

Introduction Multiple sclerosis (MS) is characterized pathologically by demyelination, axonal loss, and glial scar formation. Clinically, most patients have a relapsing-remitting course of MS (RRMS) that over time may become progressive without remissions - a secondary progressive MS (SPMS). About 15% of patients have a progressive course from onset which is called primary progressive (PP) (1). In the past decades, several treatments have been approved mainly for the use in RRMS.

Treatments for SPMS may be still effective for the early phase of this course, but it become ineffective for the later phase of SPMS (2,3) For PPMS, there is currently no approved treatment. Thus, more effective therapies need to be developed for treatment of SPMS and PPMS.

Methotrexate (MTX), an anti-metabolite, has been in clinical use since 1948 when it was found to produce temporary remission of acute childhood leukemia. Methotrexate irreversibly binds to and inhibits dihydrofolate reductase, inhibiting the formation of reduced folate, and thymidylate synthetase, resulting in inhibition of purine and thymidylic acid synthesis, thus interfering with DNA synthesis, repair, and cellular replication.

Because of its indirect immunosuppressive effects, MTX is used in treating autoimmune conditions such as rheumatoid arthritis and psoriasis (4). Low dose oral MTX (7.5 mg weekly) was found to be mildly effective, in slowing the deterioration in patients with SPMS (5).

There are accumulating evidences that in progressive MS patients there are follicular lymphoid structures in the meninges and in the Virchow-Robin spaces (8). These follicles are enriched in lymphocytes and dendritic cells which may drive the CNS inflammatory responses in the disease. This CNS restricted immune response may be unaffected by systemic immunomodulation and immunosuppressive therapies. Therefore, intrathecal therapy may target the pathological follicular lymphoid activity.

The safety of intrathecal MTX (ITMTX) has been demonstrated by its widespread use in treating lymphoproliferative diseases and leptomeningeal metastases (9). Sadik et. Al. reported about the feasibility and safety of using intrathecal methotrexate (ITMTX) as a treatment for unresponsive patients with progressive forms of MS (10). In their open label study they found that ITMTX may have a beneficial effect in progressive forms of MS and that it was well tolerated with no serious adverse events.

In the Last year the investigators have treated 8 patients with IT MTX according to the proposed protocol. Until now these patients receive 1-3 therapies of IT MTX without significance adverse event. The adverse event was were reported were: fatigue for several days post therapy and mild headache.

Objective The investigators aim is to evaluate the efficacy , safety and tolerability of intrathecal methotrexate administration in progressive MS patients.

Methods Study Population 30 progressive MS patients Inclusion Criteria

* Age 18-750 years
* Clinically definite diagnosis of MS according to McDonald criteria 2010.
* Progressive disease form defined by confirmed expanded disability status scale (EDSS) progression without relapse by at least 0.5 point or greater in the six months prior to enrollment.

Exclusion criteria

* Pregnancy
* Active infection
* Significant associated medical condition such as malignancy, heart disease or concurrent other autoimmune condition.
* Known allergy to MTX.
* WBC<4000 cells/µL
* Lym<800 cells/µL
* Treated with fingolimod or natalizumab 3 months prior to enrollment

Treatment The physician will administer 12.5 mg of MTX diluted to a concentration of up to 4 mg/mL in 0.9 percent sodium chloride with 4 mg Dexamethasone via lumbar puncture needle. These doses are standard doses of IT treatment with MTX.

Treatments will be scheduled 3 months apart for 1 year .A tota of 4 treatments in a 1 year.

A CBC with differential will be obtained before each treatment to assess the level of hematological suppression.

Evaluation A. Patients will be evaluated every 3 months by a physician other then their treating physician with the following: Kurtzke Expanded Disability Status Scale (EDSS). 25 FW , 9 PHT, Symbol Digit Modalities Test (SDMT), fatigue scale (FSS) and depression scale (BDI). In each of the visits the patient will be asked about adverse events (AE) and will be instructed to report us every AE/ medical complain he will experience between visits.

AEs will be followed until resolution or through completion of the study, whichever comes first. All Serious adverse events (SAEs) will be followed until event resolution, until the condition stabilizes, until the event is otherwise explained, or until the subject is lost to follow-up. The investigator is responsible for ensuring that follow-up includes any supplemental investigations as may be reasonably indicated to elucidate the nature and/or causality of the SAE. Any follow-up information regarding SAEs must be reported to the Helsinki committee within 24 hours.

Treatment The physician will administer 12.5 mg of MTX diluted to a concentration of up to 4 mg/mL in 0.9 percent sodium chloride with 4 mg Dexamethasone via lumbar puncture needle. These doses are standard doses of IT treatment with MTX.

Treatments will be scheduled 3 months apart for 1 year .A tota of 4 treatments in a 1 year.

A CBC with differential will be obtained before each treatment to assess the level of hematological suppression.

Laboratory test After obtaining informed consent to perform the procedure, a physician will perform a lumbar puncture with a 25 gauge needle and cerebrospinal fluid (CSF) sample will be obtained and analyze for parameters including cell count and differential, protein and glucose concentration, oligoclonal bands, IgG concentration, cellular analysis by flow cytometry for CD3+, CD20+, CD14+ cell subsets, and measurement of several soluble mediators such as: CXCL13, CD23, light chains, TNFa, IFNg, IL-17, IL-2, IL-10, BDNF and Neurofilaments will be studied by ELISA

MRI scan Brain MRI scan will be done within 1 week before each treatment. The MRI protocol includes the following sequences: T1, T2, FLAIR, T1 will gadolinium, DTI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Clinically definite diagnosis of MS according to McDonald criteria 2010.
* Progressive disease form defined by confirmed expanded disability status scale (EDSS) progression without relapse by at least 0.5 point or greater in the six months prior to enrollment.

Exclusion Criteria:

* Pregnancy
* Active infection
* Significant associated medical condition such as malignancy, heart disease or concurrent other autoimmune condition.
* Known allergy to MTX.
* WBC<4000 cells/µL
* Lym<800 cells/µL
* Treated with fingolimod or natalizumab 3 months prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The change in disability ( Multiple Sclerosis Functional Composite (MSFC) | 1 year
  Disability will be measured every visit by the Multiple Sclerosis Functional Composite (MSFC)
Safety and tolerability (adverse events) | each adverse event will be followed up until resolution
  adverse events will be followed until resolution. Serious adverse events will be reported to the IRB within 24 hours of noticed.

SECONDARY OUTCOMES:
Changes in brain MRI measurements | 1 year
  (Composite measure) We will measure new gd+ enhancing lesions, number of lesions, brain and upper spinal cord atrophy and cortical thickness and compare these measure between the time before and after treatment along. Overall each participant will undergo 5 scans , the first before treatment installation and then before each treatment . one scan will be done 3 month after the last treatment
Laboratory measurements | 1 year
  (Composite measure) Cerebrospinal fluid (CSF) sample will be obtained and analyze for parameters including cell count and differential, protein and glucose concentration, oligoclonal bands, IgG concentration, cellular analysis by flow cytometry for CD3+, CD20+, CD14+ cell subsets, and measurement of several soluble mediators such as: CXCL13, CD23, light chains, TNFa, IFNg, IL-17, IL-2, IL-10, BDNF and Neurofilaments will be studied by ELISA

REFERENCES:
- [Background] Sadiq SA (2005) Multiple sclerosis. In: Rowland LP (ed) Merritt's neurology, 11th edn. Lippincott Williams and Wilkins, Philadelphia, pp 941-963
- [Background] Goodkin DE, Rudick RA, VanderBrug Medendorp S, Daughtry MM, Schwetz KM, Fischer J, Van Dyke C. Low-dose (7.5 mg) oral methotrexate reduces the rate of progression in chronic progressive multiple sclerosis. Ann Neurol. 1995 Jan;37(1):30-40. doi: 10.1002/ana.410370108. PMID 7818255
- [Background] Hartung HP, Gonsette R, Konig N, Kwiecinski H, Guseo A, Morrissey SP, Krapf H, Zwingers T; Mitoxantrone in Multiple Sclerosis Study Group (MIMS). Mitoxantrone in progressive multiple sclerosis: a placebo-controlled, double-blind, randomised, multicentre trial. Lancet. 2002 Dec 21-28;360(9350):2018-25. doi: 10.1016/S0140-6736(02)12023-X. PMID 12504397
- [Background] American College of Rheumatology Subcommittee on Rheumatoid Arthritis Guidelines. Guidelines for the management of rheumatoid arthritis: 2002 Update. Arthritis Rheum. 2002 Feb;46(2):328-46. doi: 10.1002/art.10148. No abstract available. PMID 11840435
- [Background] Ashtari F, Savoj MR. Effects of low dose methotrexate on relapsing-remitting multiple sclerosis in comparison to Interferon beta-1alpha: A randomized controlled trial. J Res Med Sci. 2011 Apr;16(4):457-62. PMID 22091259
- [Background] Currier RD, Haerer AF, Meydrech EF. Low dose oral methotrexate treatment of multiple sclerosis: a pilot study. J Neurol Neurosurg Psychiatry. 1993 Nov;56(11):1217-8. doi: 10.1136/jnnp.56.11.1217. PMID 8229034
- [Background] Magliozzi R, Howell O, Vora A, Serafini B, Nicholas R, Puopolo M, Reynolds R, Aloisi F. Meningeal B-cell follicles in secondary progressive multiple sclerosis associate with early onset of disease and severe cortical pathology. Brain. 2007 Apr;130(Pt 4):1089-104. doi: 10.1093/brain/awm038. PMID 17438020
- [Background] Siegal T, Lossos A, Pfeffer MR. Leptomeningeal metastases: analysis of 31 patients with sustained off-therapy response following combined-modality therapy. Neurology. 1994 Aug;44(8):1463-9. doi: 10.1212/wnl.44.8.1463. PMID 8058150
- [Background] Sadiq SA, Simon EV, Puccio LM. Intrathecal methotrexate treatment in multiple sclerosis. J Neurol. 2010 Nov;257(11):1806-11. doi: 10.1007/s00415-010-5614-4. Epub 2010 Jun 10. PMID 20532907
- [Derived] Kolb H, Shachaf Y, Fainberg K, Golan M, Regev K, Vigiser I, Fuchs L, Gadoth A, Kestenbaum M, Omer N, Shopin L, Ash EL, Artzi M, Ben Bashat D, Aizenstein O, Karni A. Intrathecal methotrexate in progressive multiple sclerosis: a phase 1 open-label study with long-term follow-up. J Neurol. 2025 May 4;272(5):374. doi: 10.1007/s00415-025-13114-z. PMID 40319416